CLINICAL TRIAL: NCT05630677
Title: An Open-Label, Five-Period Study in Healthy Subjects to Investigate the Relative Bioavailability of AZD5055 Film-Coated Tablet Versus AZD5055 Oral Suspension Formulation, the Absolute Oral Bioavailability of AZD5055 and to Evaluate the Effect of Food and an Acid Reducing Agent on the Pharmacokinetics of AZD5055.
Brief Title: A Study to Compare Bioavailability of AZD5055 Film-coated Tablet With AZD5055 Oral Suspension and to Assess the Effect of Food and an Acid Reducing Agent on Pharmacokinetics (PK) of AZD5055 in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8960C00002
Record Dates: First submitted 2022-11-04; First posted 2022-11-30 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteers
Keywords: Acid Reducing Agent; Bioavailability; Healthy subjects; pH-dependent solubility; Food Effect
MeSH Terms: interventions — Rabeprazole; Tablets, Enteric-Coated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment A (Experimental): Subjects will receive AZD5055 solution as a 20-minute infusion in overnight fasted state on Day 1 in Period 1.
  Interventions: Drug: AZD5055 solution for infusion
- Treatment B (Experimental): Subjects will receive oral suspension of AZD5055 in an overnight fasted state on Day 1 in Period 1.
  Interventions: Drug: AZD5055 oral suspension
- Treatment C (Experimental): Subjects will receive AZD5055 film-coated tablet in overnight fasted state on Day 1 (Study Day 4) in Period 2.
  Interventions: Drug: AZD5055 film-coated tablet
- Treatment D (Experimental): Subjects will receive a standardized high-fat breakfast 30 minutes before film-coated tablet of AZD5055 administered as On Day 1 (Study Day 8) in Period 3.
  Interventions: Drug: AZD5055 film-coated tablet
- Treatment E (Experimental): Subjects will receive rabeprazole twice daily on Day 10. On Day 1 (Study Day 13), AZD5055 film-coated tablet will be administered, under fasted conditions, together with rabeprazole and rabeprazole dosing will continue twice daily in Period 4.
  Interventions: Drug: AZD5055 film-coated tablet; Drug: Rabeprazole, Delayed-release tablet
- Treatment F (Experimental): Subjects will receive a low-fat breakfast 30 minutes before AZD5055 film-coated tablet administered together with rabeprazole on Day 17. Rabeprazole will continue twice daily, the last dose is on the evening of Study Day 18 in Period 5.
  Interventions: Drug: AZD5055 film-coated tablet; Drug: Rabeprazole, Delayed-release tablet

INTERVENTIONS:
Drug: AZD5055 solution for infusion — Subjects will receive a single dose intravenous infusion of AZD5055 as 20-minute infusion on Day 1 of the respective period in overnight fasted state.
  Arms: Treatment A
Drug: AZD5055 oral suspension — Subjects will receive single dose of AZD5055 oral suspension on Day 1 of the respective period in overnight fasted state.
  Arms: Treatment B
Drug: AZD5055 film-coated tablet — Subjects will receive single oral dose of AZD5055 film-coated tablets on Day 1 of the respective period in overnight fasted state.
  Arms: Treatment C; Treatment E
Drug: AZD5055 film-coated tablet — Subjects will receive single oral dose of AZD5055 film-coated tablets on Day 1 of the respective period in fed state (either a high fat meal or low-fat meal calorie standard breakfast)
  Arms: Treatment D; Treatment F
Drug: Rabeprazole, Delayed-release tablet — Subjects will receive oral doses of rabeprazole twice daily 3 days prior to AZD5055 single dose and 4 days after the AZD5055 single dose including the day that AZD5055 is dosed under fasted conditions [Study Day 10 to 18].
  Arms: Treatment E
Drug: Rabeprazole, Delayed-release tablet — Subjects will receive oral doses of rabeprazole twice daily prior to AZD5055 single dose under fed conditions (low-fat standard breakfast) and then continued for 2 days.
  Arms: Treatment F

SUMMARY:
This study will estimate the relative bioavailability of AZD5055 film-coated tablet as compared to AZD5055 oral suspension. The study will also assess the absolute bioavailabilty of AZD5055 and the effect of food and an acid reducing agent, rabeprazole, on the PK of AZD5055 film-coated tablets when given with food (fed state) or without food (fasted state).

DETAILED DESCRIPTION:
This will be an Open-Label, Five-Period Study in healthy subjects. The study will comprise of a Screening Period of maximum 28 days.

The treatment groups are as follows:

* Treatment A: AZD5055 solution for infusion as 20-minute infusion and an overnight fasted state after the 20-minute infusion.
* Treatment B: AZD5055 oral suspension and an overnight fasted state after the oral suspension.
* Treatment C: AZD5055 film-coated tablet and an overnight fasted state after the film-coated tablet..
* Treatment D: AZD5055 film-coated tablet, fed state (after a high-fat, high-calorie standard breakfast).
* Treatment E: Twice daily oral doses of 20 mg rabeprazole for 3 days prior a single dose of AZD5055 film-coated tablet under fasted conditions, and then rabeprazole will be continued for 2 days.
* Treatment F: Twice daily oral doses of 20 mg rabeprazole continuing from Treatment E prior to a single dose of AZD5055 film-coated tablet under fed conditions (low-fat standard breakfast) and then rabeprazole will be continued for 2 days.

Five (5) periods during which subjects will participate from Day -1 of Period 1 to 72 hours after the AZD5055 dose in Period 5.

* Period 1: On Day 1, the subjects will receive either Treatment A or Treatment B.
* Period 2: On Day 4, the subjects will receive Treatment C.
* Period 3: On Day 8, the subjects will receiveTreatment D.
* Period 4: On Day 10, three days prior to Day 1, rabeprazole will be administered twice daily. On Day 13, subject will receive Treatment E.
* Period 5: On Day 17, the subjects will receive Treatment F. Rabeprazole will continue twice daily, the last dose is on the evening of Study Day 18.

A Follow-up Visit, or telephone call, approximately 6 days after the last AZD5055 dose in Period 5.

There will be a minimum washout of 3 days between the AZD5055 dose administration in Period 1 and Period 2 and a minimum washout of 4 days between AZD5055 doses administrations for subsequent study periods.

Each subject will participate in the study for approximately 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female (of non-childbearing potential) subjects aged 18 to 55 years.
2. Female subjects must have a negative pregnancy test.
3. Male subjects must adhere to the contraception methods as per Protocol.
4. Have a BMI between 18 and 30 kg/m2 inclusive.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which may either put the subject at risk because of participation in the study or influence the results or the subject's ability to participate in the study.
2. Ongoing acute Gastrointestinal (GI), hepatic, or renal disease, a history of chronic GI, hepatic, or renal disease, pancreatic disease, diabetes mellitus, or any condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study drug.
4. Ongoing acquired or inherited immunodeficiency disorders, including but not limited to Human Immunodeficiency Virus (HIV) or common variable immunodeficiency, or the subject is taking immune replacement therapy.
5. Individuals with chronic infections or who are at increased risk of infection.
6. History of cancer within the last 10 years (20 years for breast cancer). Any history of lymphoma is not allowed.
7. History of osteoporosis, osteomalacia, Paget's disease of the bone, thyrotoxicosis, rheumatoid arthritis, Cushing's disease, or a pathological fracture.
8. History of a traumatic fracture within 6 months of the Screening Visit.
9. Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis.
10. Abnormal vital signs. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG and any clinically important abnormalities in the 12-lead ECG.
11. Untreated tuberculosis (TB) or a positive result for the Interferon gamma release assay (IGRA) (ie, QuantiFERON TB Gold).
12. Any positive result at Screening for serum hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C antibody, and HIV antibody.
13. History of severe COVID-19 infection requiring hospitalization within the last 12 months prior to Screening, or clinical history compatible with Long COVID-19 (symptoms beyond 12 weeks of acute infection).
14. Confirmed COVID-19 infection during at admission.
15. Has received live or live attenuated vaccine in the 30 days prior to dosing, the first dose of COVID- vaccine within 30 days prior to randomization, or a COVID-19 vaccine second or booster vaccination within 10 days of Screening.
16. Known or suspected history of drug abuse.
17. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity.
18. Current smokers or use of any tobacco in any other form.
19. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol.
20. Use of drugs with enzyme-inducing properties such as St John's Wort.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Area under concentration time curve from time 0 to infinity (AUCinf) | Day 1-6, 8-10, 13-15, 17-19
  * To estimate the relative bioavailability of AZD5055 film-coated tablet formulation versus AZD5055 oral suspension formulation.
  * To estimate the absolute bioavailability of AZD5055 oral suspension and AZD5055 film-coated tablet formulation.
  * To assess the effect of the acid reducing agent, rabeprazole, on the PK of AZD5055 alone and in combination with acid reducing agent.
  * To assess the effect of the acid reducing agent, rabeprazole, on the PK of AZD5055, when AZD5055 is administered.
Area under the concentration time curve from time 0 to the last quantifiable concentration (AUClast) | Day 1-6, 8-10, 13-15, 17-19
  * To estimate the relative bioavailability of AZD5055 film-coated tablet formulation versus AZD5055 oral suspension formulation.
  * To estimate the absolute bioavailability of AZD5055 oral suspension and AZD5055 film-coated tablet formulation.
  * To assess the effect of food on the pharmacokinetic (PK) parameters of AZD5055 in the fed and fasted state.
  * To assess the effect of the acid reducing agent, rabeprazole, on the PK of AZD5055 alone and in combination with acid reducing agent.
  * To assess the effect of the acid reducing agent, rabeprazole, on the PK of AZD5055, when AZD5055 is administered in fasted and fed state.
Maximum observed concentration (Cmax) | Day 1-6, 8-10, 13-15, 17-19
  * To estimate the relative bioavailability of AZD5055 film-coated tablet formulation versus AZD5055 oral suspension formulation.
  * To estimate the absolute bioavailability of AZD5055 oral suspension and AZD5055 film-coated tablet formulation.
  * To assess the effect of food on the pharmacokinetic (PK) parameters of AZD5055 in the fed and fasted state.
  * To assess the effect of the acid reducing agent, rabeprazole, on the PK of AZD5055 alone and in combination with acid reducing agent.
  * To assess the effect of the acid reducing agent, rabeprazole, on the PK of AZD5055, when AZD5055 is administered in fasted and fed state.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, MD, Principal Investigator — PAREXEL Early Phase Clinical Unit Baltimore
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: D8960C00002_CSR Synopsis_Redacted.pdf — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8960C00002&attachmentIdentifier=cd60401e-c3ff-4505-bbd5-a71f8f695602&fileName=D8960C00002_CSR_Synopsis_Redacted.pdf&versionIdentifier=